CLINICAL TRIAL: NCT06086340
Title: Comparative Assessment of Overall Survival in Medicare Patients With HR+/HER2- Metastatic Breast Cancer Treated With Palbociclib in Combination With Aromatase Inhibitor (AI vs. AI Alone)
Brief Title: Study to Compare Overall Survival in Medicare Patients With Metastatic Breast Cancer Treated With a Medicine Called Palbociclib in Combination With Aromatase Inhibitor and Aromatase Inhibitor by Itself.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481182; Henri 3 (Other: Alias Study Number)
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Breast neoplasm; Hormone receptor-positive Human epidermal growth factor receptor 2 negative (HR+,HER2-); palbociclib; Metastatic; Medicare; SEER-Medicare
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — palbociclib; Aromatase Inhibitors; Letrozole; Anastrozole; exemestane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Palbociclib + AI: Adult metastatic breast cancer patients who initiated Palbociclib + an aromatase inhibitor as first line therapy in SEER-Medicare
  Interventions: Drug: Palbociclib; Drug: Aromatase Inhibitor
- AI alone: Adult metastatic breast cancer patients who initiated an aromatase inhibitor (alone) as first line therapy
  Interventions: Drug: Aromatase Inhibitor

INTERVENTIONS:
Drug: Palbociclib — Palbociclib with an aromatase inhibitor therapy
  Other Names: Ibrance
  Groups: Palbociclib + AI
Drug: Aromatase Inhibitor — Aromatase Inhibitor Therapy
  Other Names: letrozole, anastrozole, exemestane

SUMMARY:
A retrospective study of de-identified (to preserve patient privacy) patient information from the SEER-Medicare Database to compare overall survival of first line palbociclib + aromatase inhibitor (AI) therapy versus AI therapy alone treatment in women or men aged 65 and older with newly diagnosed hormone receptor positive/human epidermal growth factor receptor 2 negative (HR+/HER2-) metastatic breast cancer (MBC) in the United States

ELIGIBILITY:
Inclusion Criteria:

* De novo metastatic (stage IV) disease at initial breast cancer diagnosis during 2015-2019
* HR+/HER2- molecular subtype at diagnosis
* Initiated 1L systemic therapy with palbociclib + AI or AI alone

Exclusion Criteria:

* Patients will be excluded if their metastatic breast cancer diagnosis was first recorded in a death certificate or at the time of autopsy.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Medicare recipients with HR+/HER2- with De Novo metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 779 (Actual)
Dates: Start 2023-09-29 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Brufsky AM, Sandin R, Stergiopoulos S, Chen C, Karanth S, Li B, Esterberg E, Makari D, Candrilli SD, Goyal RK, Rugo HS. Overall Survival With Palbociclib and Aromatase Inhibitor Versus Aromatase Inhibitor Alone in Older Patients With HR+/HER2- Metastatic Breast Cancer. Cancer Med. 2025 Apr;14(7):e70719. doi: 10.1002/cam4.70719. PMID 40145289
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481182

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of eligible participants diagnosed with hormone receptor (HR+)/ human epidermal growth factor receptor 2-negative (HER2) metastatic breast cancer (mBC) treated with palbociclib in combination with aromatase inhibitor (AI) was extracted from clinical and administrative claims data from the linked surveillance, epidemiology, and end results (SEER)-Medicare database from 1-August-2014 until 31-December-2020 were observed retrospectively.
Pre-assignment Details: Available data from eligible participants was evaluated in approximately 4 months of this retrospective observational study.
Groups:
- AI Alone: Participants who received an AI (alone) as first line therapy under standard real world routine clinical practice for HR+/HER2- mBC during the period 1-February-2015 to 30-June-2020 were included in this retrospective observational study.
- Palbociclib + AI: Participants who received Palbociclib in combination with an AI under standard real world routine clinical practice for HR+/HER2- mBC during the period 1-February-2015 to 30-June-2020 were included in this retrospective observational study.
Period: Overall Study
Arm/Group | AI Alone | Palbociclib + AI
Started | 483 | 296
Completed | 483 | 296
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data was extracted and evaluated for the retrospective analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | AI Alone | Palbociclib + AI | Total
Number analyzed (Participants) | 483 | 296 | 779
Age, Customized [Count of Participants; unit: Participants]
  65-69 years | 86 | 86 | 172
  70-74 years | 91 | 84 | 175
  75-79 years | 101 | 67 | 168
  Greater than or equal to (>=) 80 years | 205 | 59 | 264
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Here "number analyzed" signifies participant evaluable for this baseline measure.
  Participants
    number analyzed (Participants) | 480 | 294 | 774
    Female | 480 | 294 | 774
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 14 | 37
  Not Hispanic or Latino | 460 | 282 | 742
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Here "number analyzed" signifies participant evaluable for this baseline measure.
  Participants
    Race: number analyzed (Participants) | 476 | 292 | 768
    Race: American Indian or Alaska Native | 0 | 0 | 0
    Race: Asian or Pacific Islander | 14 | 13 | 27
    Race: Black | 45 | 23 | 68
    Race: White | 417 | 256 | 673
    Race: Other or unknown | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival According to Unadjusted Analysis
Description: Overall survival was defined as time in months from the study index date to all cause death. Study index date in this outcome measure was the date of first line of treatment initiation with palbociclib + AI or AI alone after the de novo mBC diagnosis. De novo mBC referred to breast cancer that physician diagnosed for the first time after it had already spread outside of the breast to distant parts of the body. Unadjusted analysis: analysis not considering any covariates, specifically potential differences in baseline characteristics that could confound the association between treatment and survival. Overall survival was assessed using Kaplan-Meier analysis.
Time Frame: From index date to death (approximately 69.9 months); retrospective data evaluated in 4 months (approximately) of this study
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AI Alone | Palbociclib + AI
Number analyzed (Participants) | 483 | 296
Months | 24.2 [20.5 to 26.7] | 44.0 [37.3 to 54.5]

2. Primary Outcome: Overall Survival According to Stabilized Inverse Probability of Treatment Weighted (sIPTW) Analysis
Description: Overall survival was defined as time in months from the study index date to all cause death. Study index date in this outcome measure was the date of first line of treatment initiation with palbociclib + AI or AI alone after the de novo mBC diagnosis. De novo mBC referred to breast cancer that physician diagnosed for the first time after it had already spread outside of the breast to distant parts of the body. sIPTW analysis: stabilized inverse probability treatment weighting. This is a statistical method that reweights participants to create groups with similar baseline characteristics. The analysis therefore adjusts for differences in baseline characteristics that could confound the association between treatment and survival. Overall survival was assessed using Kaplan-Meier analysis.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AI Alone | Palbociclib + AI
Number analyzed (Participants) | 483 | 296
Months | 25.5 [22.0 to 28.9] | 37.6 [34.8 to 42.0]

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored; hence time frame is not applicable. For all-cause mortality: from index date to death (approximately 69.9 months); retrospective data evaluated in 4 months (approximately) of this study
Description: Due to non-interventional nature of study, the minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) were not met, hence adverse events were not monitored. Thus, participants at risk are zero for adverse events.
Arm/Group | AI Alone | Palbociclib + AI
All-Cause Mortality (participants affected / at risk) | 279/483 | 113/296
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT06086340/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT06086340/SAP_001.pdf